CLINICAL TRIAL: NCT07214272
Title: A Phase 4 Clinical Study to Investigate the Effectiveness and Safety of Skin Resurfacing Procedures Using the Next Generation Fraxel® FTX Laser System in Participants With Dyschromia, Cutaneous Lesions, and Periorbital Rhytids
Brief Title: A Phase 4 Clinical Study to Investigate the Effectiveness and Safety of Skin Resurfacing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX-PAS-USA-2024-001
Record Dates: First submitted 2025-09-18; First posted 2025-10-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Skin Resurfacing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: Fraxel® FTX Laser System

INTERVENTIONS:
Device: Fraxel® FTX Laser System — The Fraxel Laser System has two fiber-laser sources that are contained in a single Console. The Console is electrically connected to the facility power source. Laser energy produced by the unit is delivered to the tissue through the Handpiece, which is connected to the Console by the Handpiece Cable. Treatments are delivered through removable, disposable Treatment Tips which attach to the Handpiece. A Treatment Key is required to activate treatments and is inserted into the port on the side of the Touchscreen.
  The system includes two lasers with wavelengths of 1550 nm and 1927 nm. The two-wavelength option allows for targeted treatment of different tissue depths, and the wavelength can be selected through the Console Touchscreen. Interchangeable Tips allow for treatment of both small and large areas.

SUMMARY:
This study is a prospective, post-marketing (Phase 4) non-registrational single-arm, open-label, multicenter study.

DETAILED DESCRIPTION:
Study to be conducted at approximately 6 investigative sites in the United States, enrolling up to 50 male and female participants with Fitzpatrick skin types I to VI, with no more 30 (60%) participants with Fitzpatrick skin types I to III and approximately 20 (40%) participants who self-identify as being of Asian descent

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. 21 to 60 years of age.
3. Written informed consent must be obtained prior to any study procedures.
4. Presence of one or more of the following in the treatment area(s):

   1. Photodamage as determined by investigator using a Modified Griffith's Scale (score of 3 to 7 in overall photodamage on the 9-point scale)
   2. Mild-to-moderate rhytids (e.g., periorbital crow's feet) as determined by investigator using a Modified Griffith's Scale (score of 3 to 6 on the 9-point scale).
   3. Mild-to-severe dyschromia, including lentigos or solar lentigines as determined by investigator using the Modified Griffith's Scale (score of 3 to 9 on the 9-point scale).
5. Ability to read, understand, and sign the informed consent form

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant during the study.
2. History of any type of allergic reaction to topical anesthetics.
3. Localized infection in the treatment area or systemic infection within the last 1 month prior to or at any time during the study.
4. Presence of melasma, rosacea, significant actinic keratoses, or other significant skin conditions in the target treatment zone.
5. Presence of skin cancer, infection, cold sore, open wounds, burns, psoriasis, or active dermatitis of any kind (atopic, contact, significant seborrheic dermatitis) in the target treatment zone.
6. Presence of skin conditions that, in the judgement of the investigator, would increase the risk of study participation or treatment.
7. Predisposition to keloid formation or excessive scarring.
8. Diagnosis of a condition that may compromise the immune system, such as: HIV, lupus, and/or scleroderma.
9. Known sensitivity to light or photosensitizing agents/medications are being taken that the investigator determines may affect study treatment.
10. Use of systemic steroids (e.g. prednisone, dexamethasone) or other immunosuppressants within 1 month prior to enrollment to or at any time during the study.
11. Use of topical retinoids within 2 weeks prior to enrollment or at any time during the study.
12. Use of systemic retinoids within 6 months prior to enrollment or at any time during the study.
13. Had a cosmetic procedure, such as a chemical peel, mechanical peel, laser resurfacing, and/or skin tightening procedures (microneedling, ultrasound, etc.) within the previous 4 months prior to enrollment.
14. Receiving short-acting botulinum toxin within 4 months or long-acting botulinum toxin administered to the targeted treatment zone within 9 months prior to enrollment or at any time during the study.
15. Receiving dermal fillers administered to the targeted treatment zone within 3 months prior to enrollment or at any time during the study.
16. Sunburn and/or significant recent sun exposure on the target treatment zone in the last 2 weeks prior to enrollment that, according to investigator judgement, would impact treatment, and/or unwilling to practice photoprotection and/or avoid significant sun exposure for the duration of study participation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 26 weeks
  Proportion of participants with any improvement after 3 treatments as assessed by Investigator Global Aesthetic Improvement Scale (iGAIS) at End of Study

SECONDARY OUTCOMES:
Secondary Endpoint | 26 weeks
  The FACE-Q Satisfaction with Outcome domain will be administered at the EOS visit to evaluate participant-reported satisfaction following Fraxel FTX treatments.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dermatology Cosmetic Laser Associates of La Jolla, Inc. d/b/a West Dermatology Research Center, La Jolla, California
  - Miami Dermatology & Laser Research LLC, Miami, Florida
  - Oak Dermatology, LLC, Naperville, Illinois
  - Union Square Laser Dermatology, P.C, New York, New York
  - Dermatology and Laser Surgery Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No